CLINICAL TRIAL: NCT01032863
Title: A Study of Association Between Hypermobility And Chronic MusculoSkeletal Pain:a Pilot Study
Brief Title: Association Between Hypermobility and Chronic Musculoskeletal Pain
Acronym: HAMS
Status: Completed | Type: Observational
Sponsor: Amrita Institute of Medical Sciences & Research Center (Other)
Responsible Party: Sharath Kumar, Amrita Institute of Medical Sciences
Other Study IDs: K-PAE-09-258
Record Dates: First submitted 2009-12-14; First posted 2009-12-16 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2009-12

CONDITIONS: Hypermobility, Joint; Arthralgia; Myofascial Pain Syndromes; Fibromyalgia; Pain Disorder
Keywords: Chronic musculoskeletal pain; Benign joint hypermobility syndrome; Fibromyalgia
MeSH Terms: conditions — Joint Instability; Arthralgia; Myofascial Pain Syndromes; Fibromyalgia; Somatoform Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Young healthy Indian adults: Persons aged between 25 and 40 years of age who are relatives of patients being treated in Amrita Institute of Medical Sciences (Inpatient or Outpatient) and voluntary blood donors at the same institute who are willing to participate in the study.

SUMMARY:
Study hypothesis:- Benign joint hyper mobility syndrome which persists into adulthood is a special type of benign joint hyper mobility which is more likely to predispose to chronic musculoskeletal pain.

Young Indian adults aged between 25 and 40 years who are blood donors or relatives of patients admitted as inpatient or presenting to the out patient department, in Amrita Institute of Medical Sciences will be enrolled, after excluding the exclusionary criteria. They will be assessed for the presence of chronic musculoskeletal pain using a validated self filled questionnaire. The primary investigator who will be blinded to their response will examine them for the presence of Benign Joint Hyper mobility Syndrome and for tender points suggestive of fibromyalgia.

Primary Objective:- To determine whether chronic musculoskeletal pain is associated with Hypermobility among Indian adults.

Study design:- Cross sectional survey

ELIGIBILITY:
Inclusion Criteria:

1. Completed their 25th birthday
2. Not yet celebrated their 40th birthday
3. Are relatives of patients being treated in Amrita Institute of Medical Sciences or voluntary blood donors in the same institute

Exclusion Criteria:

1. Subjects who have been diagnosed previously with a inflammatory musculoskeletal disease.
2. Subjects detected to have signs or symptoms of inflammatory arthritis on a detailed clinical examination and history taking.
3. Subjects who have symptoms suggestive of diabetes mellitus or hypothyroidism or have been previously diagnosed with the same.
4. Subjects who are not willing to participate.
5. Subjects who have been diagnosed as having a connective tissue disorder or have a family history of the same.

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Young Indian adults aged between 25 years and 40 years
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2009-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
To determine whether chronic musculoskeletal pain is associated with hypermobility among young Indian adults | 3-6 months

SECONDARY OUTCOMES:
Determine whether hypermobility is associated with the presence of fibromyalgia in young Indian adults. | 3-6 months
Determine the prevalence of hypermobility among Indian adults | 3-6 months
Determine prevalence of fibromyalgia in young Indian adults | 3-6 months
Determine the prevalence of chronic musculoskeletal pain among young indian adults | 3-6 months
Determine the association between American College of Rheumatology criteria for definition of Fibromyalgia and Simplified intensity scale questionnaire definition of Fibromyalgia. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sharath Kumar, MD, Principal Investigator — Amrita Institute of Medical Sciences; L Rajam, MD, Study Director — Amrita Institute of Medical Sciences
Locations (1):
- Amrita Institute of Medical Sciences, Kochi, Kerala, India

REFERENCES:
- [Background] Leone V, Tornese G, Zerial M, Locatelli C, Ciambra R, Bensa M, Pocecco M. Joint hypermobility and its relationship to musculoskeletal pain in schoolchildren: a cross-sectional study. Arch Dis Child. 2009 Aug;94(8):627-32. doi: 10.1136/adc.2008.150839. Epub 2009 May 12. PMID 19465584
- [Background] Mikkelsson M, Salminen JJ, Kautiainen H. Joint hypermobility is not a contributing factor to musculoskeletal pain in pre-adolescents. J Rheumatol. 1996 Nov;23(11):1963-7. PMID 8923376
- [Background] Engelbert RH, Bank RA, Sakkers RJ, Helders PJ, Beemer FA, Uiterwaal CS. Pediatric generalized joint hypermobility with and without musculoskeletal complaints: a localized or systemic disorder? Pediatrics. 2003 Mar;111(3):e248-54. doi: 10.1542/peds.111.3.e248. PMID 12612280
- [Background] Sendur OF, Gurer G, Bozbas GT. The frequency of hypermobility and its relationship with clinical findings of fibromyalgia patients. Clin Rheumatol. 2007 Apr;26(4):485-7. doi: 10.1007/s10067-006-0304-4. Epub 2006 Apr 25. PMID 16636935